CLINICAL TRIAL: NCT03392675
Title: Promoting Self-Management of Breast and Nipple Pain in Breastfeeding Women
Brief Title: Breastfeeding Self-Management for Nipple and Breast Pain
Acronym: BSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H16-321; 5P20NR016605-02 (NIH)
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Breastfeeding; Breast Pain
Keywords: Breast and Nipple Pain; Quantitative Sensory Testing; Genotyping; Breastfeeding
MeSH Terms: conditions — Breast Feeding; Mastodynia | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Masking Description: Using a stratified and blocked randomization scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-monitoring of BF and intervention (Experimental): Self-monitoring and regulation skills will be provided to mothers at discharge. Aside from daily diaries outlining, infant feeding behaviors and pain, mothers will be instructed to watch several 5-minute video modules to assist with self-management of breast and nipple pain. These videos include: pain neurophysiology; non-pharmacological strategies; common BF issues and intervention; catastrophizing; stress reactivity; deep breathing; guided imagery and support (informational and instrumental). These mothers will also be asked to complete study questionnaires and measures at specified time points.
  Interventions: Behavioral: Self-monitoring of BF and intervention
- Control (No Intervention): Usual care and asked to complete measures at follow-up time points.

INTERVENTIONS:
Behavioral: Self-monitoring of BF and intervention — Self-Monitoring: At discharge, mothers will complete daily diaries for self-monitoring to stimulate cognitive reframing on the occurrence, duration, and characteristics of nipple and breast pain, infants' latch and sucking pattern, positioning, length of each BF session, and the MAIBB.
  Self-Regulation: To support self-regulation skills, mothers will be provided with several 5-minute video modules on pain and BF pain SM with additional resources links. After discharge mother will receive text message from a nurse 2X/week for BF support. Mothers may text the nurse for emergent BF support.
  Arms: Self-monitoring of BF and intervention

SUMMARY:
This pilot project will provide an understanding of the contextual variables responsible for breast and nipple pain during breastfeeding initiation. These variables include, genetic variation, pain sensitivity, reactivity, pain catastrophizing and perceived stress. The purpose is to understand the efficacy of self-management (SM) strategies on each of these contextual variables, in an effort to inform a personalized approach to managing breastfeeding pain and its effect on improved health outcomes.

DETAILED DESCRIPTION:
Breastfeeding (BF) is one of the most important early determinants of infant health and development. Duration of BF is significantly related to reduced incidence of infantile respiratory and gastrointestinal tract infections, obesity and asthma. However, over 35% of mothers cease exclusive BF during the first 6 weeks due to nipple and breast pain. While 90% of mothers report acute nipple and breast pain during the first week of BF initiation, approximately 30% will experience persistent pain (>10 days). Due to the significant impact of nipple and breast pain on BF duration, pain is a significant barrier for achieving public health outcomes.

The following pilot project will test the feasibility of a Breastfeeding Self-Management (BSM) Intervention on BF outcomes in mothers with nipple and breast pain. In addition, the proposed study will provide a preliminary examination of genetic, psychological and somatosensory factors that predict nipple and breast pain and possibly, early cessation of BF.

Individual factors, including genetic polymorphisms of pain sensitivity genes and the individual's interpretation of pain can influence pain facilitation or inhibition at the molecular level of pain processing. Moreover, maternal anticipation of pain may increase pain catastrophizing, perceived stress and reactivity contributing to increased peripheral and central sensitivity. Identifying strategies to increase mothers' BF knowledge, pain self-efficacy and self-regulation skills could lead to increased SM behaviors. Therefore, this pilot study was designed to target pain SM process factors (self-monitoring, knowledge of breast care, BF self-efficacy, pain self-efficacy, and problem solving) relevant to mothers who experience pain during BF. The overarching goal of this program of research is to improve nipple and breast pain SM in BF mothers and enhance their BF self-efficacy to achieve their BF goals.

The proposed study will address a major barrier of BF duration by identifying factors that contribute to nipple and breast pain. The proposed SM intervention will specifically target pain information, pain self-efficacy and problem-solving as central components of the SM process. In addition, the investigators will examine the influence of peripheral and central sensitivity and frequency of catechol-O-methyltransferase (COMT) single-nucleotide polymorphisms (SNPs), on SM process and outcome variables over time to gain knowledge about the precise influence of the molecular context of pain on risk of nipple and breast pain and BF outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have just given birth (<48 hours)
* Intention to breastfeed for 6 weeks
* Has daily access to a computer with internet
* Access to a phone
* Read and speak English
* Delivered a healthy singleton infant born >37 weeks gestational age

Exclusion Criteria:

* Infants with congenital anomalies
* Mothers with major mental health issues (i.e Schizophrenia, Mania, Bipolar Disorder)
* Complications during delivery requiring intervention
* Mothers with major health issues that are not associated with pregnancy as determined by principal investigator (i.e. infection illness such as HIV+, hepatitis, diabetes, history of seizures, current diagnosis of cancer).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Pain Sensitivity | Baseline
  Quantitative sensory testing
Genetic variations in COMT | Baseline
  Pain susceptibility SNPs genotyping related to breastfeeding related breast and nipple pain.

SECONDARY OUTCOMES:
Increased duration of breastfeeding | Week 1, 2 and 6
  With self-management of breast and nipple pain

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Lucas, PhD, RN, Principal Investigator — University of Connecticut
Locations (2):
- United States (2):
  - UConn Health, Farmington, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that are part of National Institute of Nursing Research (NINR) designated common data elements collected during the trial, after de-identification have been submitted to NIH repository at the Common Data Repository for Nursing Science (cdRNS). Data can be accessed by directly submitting requests at that website.
  When will data be available (start and end dates)? Immediately. No end date.
  With whom? Anyone who wishes to access the data and creates an account on cdRNS.nih.gov.
  By what mechanism will data be made available? Data are available at cdRNS.nih.gov
Time Frame: within 2 years
Access Criteria: Requests will be submitted through the cdRNS website.

REFERENCES:
- [Background] Breastfeeding. J Obstet Gynecol Neonatal Nurs. 2015 Jan-Feb;44(1):145-50. doi: 10.1111/1552-6909.12530. Epub 2015 Jan 14. No abstract available. PMID 25588888
- [Background] Odom EC, Li R, Scanlon KS, Perrine CG, Grummer-Strawn L. Reasons for earlier than desired cessation of breastfeeding. Pediatrics. 2013 Mar;131(3):e726-32. doi: 10.1542/peds.2012-1295. Epub 2013 Feb 18. PMID 23420922
- [Background] Kent JC, Ashton E, Hardwick CM, Rowan MK, Chia ES, Fairclough KA, Menon LL, Scott C, Mather-McCaw G, Navarro K, Geddes DT. Nipple Pain in Breastfeeding Mothers: Incidence, Causes and Treatments. Int J Environ Res Public Health. 2015 Sep 29;12(10):12247-63. doi: 10.3390/ijerph121012247. PMID 26426034
- [Background] Dennis CL, Jackson K, Watson J. Interventions for treating painful nipples among breastfeeding women. Cochrane Database Syst Rev. 2014 Dec 15;2014(12):CD007366. doi: 10.1002/14651858.CD007366.pub2. PMID 25506813
- [Background] Nicholas Penney, J., The biopsychosocial model of pain and contemporary osteopathic practice. International Journal of Osteopathic Medicine, 2010. 13(2): p. 42---47.
- [Background] Amir LH, Jones LE, Buck ML. Nipple pain associated with breastfeeding: incorporating current neurophysiology into clinical reasoning. Aust Fam Physician. 2015 Mar;44(3):127-32. PMID 25770578
- [Background] Diatchenko L, Slade GD, Nackley AG, Bhalang K, Sigurdsson A, Belfer I, Goldman D, Xu K, Shabalina SA, Shagin D, Max MB, Makarov SS, Maixner W. Genetic basis for individual variations in pain perception and the development of a chronic pain condition. Hum Mol Genet. 2005 Jan 1;14(1):135-43. doi: 10.1093/hmg/ddi013. Epub 2004 Nov 10. PMID 15537663
- [Derived] Lucas R, Zhang Y, Walsh SJ, Evans H, Young E, Starkweather A. Efficacy of a Breastfeeding Pain Self-Management Intervention: A Pilot Randomized Controlled Trial. Nurs Res. 2019 Mar/Apr;68(2):E1-E10. doi: 10.1097/NNR.0000000000000336. PMID 30829925
- See also: Center for Accelerating Precision Pain Self-Management (CAPPS-M) Website — https://cappsm.nursing.uconn.edu/

DOCUMENTS (1):
  • Informed Consent Form (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT03392675/ICF_000.pdf